CLINICAL TRIAL: NCT06005649
Title: A Multi-center, Open Label, Single-arm, Phase I/II Clinical Trial of HY004 Cell Injection in the Treatment of Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma
Brief Title: Clinical Trial of HY004 Cell Injection in the Treatment of Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor changed product development plan
Sponsor: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY004102
Record Dates: First submitted 2023-08-17; First posted 2023-08-22 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Non-hodgkin Lymphoma
Keywords: HY004; CD22/CD19 Chimeric Antigen Receptor T-cells
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single dose of HY004 (Experimental): Patients received a single dose of anti-CD22/CD19 CAR T cells after receiving a conditioning regimen of cyclophosphamide and fludarabine.
  Interventions: Biological: HY004

INTERVENTIONS:
Biological: HY004 — Autologous 2nd generation bispecific CAR-T cells targeting both CD22 and CD19, single infusion intravenously.
  Start Dose level: 2.00 x 10^6/kg CAR+T-cells

SUMMARY:
This is a multi-center, open-label, single-arm, phase I/II trial to evaluate the safety and efficacy of HY004 treatment in Adult patients with relapsed or refractory B-cell Non-Hodgkin's Lymphoma (r/r B-NHL).

DETAILED DESCRIPTION:
This trial is a multi-center, open label, single-arm, phase I/II trial to evaluate the safety and efficacy of HY004 in Adult(aged 18~75 years old) patients with r/r B-NHL.

The phase I part of the trial is to evaluate the safety, optimal dose of HY004, Pharmacokinetics/Pharmacodynamics(PK/PD)and preliminary efficacy in the treatment of Adult patients with r/r B-NHL. The phase II part of the trial is to evaluate the efficacy and safety of HY004 in in the treatment of Adult patients with r/r B-NHL. The study includes screening, pre-treatment (Cell Product manufacture & lymphodepletion), HY004 infusion , safety and efficacy follow-up, and survival follow-up. All subjects who have received HY004 infusion will be followed for up to 2 years.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients who are willing to sign the informed consent form;
2. Aged 18-75 years, male or female;
3. Previously received≥2nd-line adequate therapy or hematopoietic stem cell transplantation (HSCT), and patients with CD19+/CD22+ relapsed/refractory B-NHL according to the WHO classification 2017, which are provided specifically as follows:

   1. Diffuse large B cell lymphoma (DLBCL), not otherwise specified (NOS);
   2. Primary mediastinal large B cell lymphoma (PMBCL);
   3. Grade 3b follicular lymphoma;
   4. Transformed follicular lymphoma;
   5. High grade B cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements, and high grade B cell lymphoma - not otherwise specified.
4. Measurable imaging lesion at screening: Intranodal lesion must have a long diameter of more than 1.5 cm, and extranodal lesion must have a long diameter of more than 1.0 cm with PET-positive disease by Lugano classification .
5. PET-positive disease BY Lugano classification
6. Adequate bone marrow, renal, hepatic, pulmonary and cardiac function.
7. Adequate vascular access for leukapheresis procedure
8. Subjects who have received previous CD19-targeted therapy must have CD19-positive lymphoma confirmed on a biopsy since completing the prior CD19-targeted therapy.

Key Exclusion Criteria:

1. Active Central Nervous System (CNS) involvement by malignancy.
2. Patients with existing central nervous system disease or with a history of central nervous system disease.
3. Patients receiving any of the following drugs or therapies within the specified period prior to apheresis:

   1. Alemtuzumab and Bendamustine within 6 months prior to apheresis;
   2. Cladribine within 3 months prior to apheresis;
   3. Lenalidomide within 1 mouth prior to apheresis;
   4. Lymphocytotoxic chemotherapy within 2 weeks prior to apheresis - use in more than 3 half-lives prior to apheresis is eligible;
   5. Anti-CD20 monoclonal antibody and therapeutic dose of hormones within 7 d prior to apheresis;
   6. Non-lymphocytotoxic chemotherapy within 7 d prior to apheresis - use in more than 3 half-lives prior to apheresis is eligible;
   7. Venetoclax (BCL-2 inhibitor) within 4 d prior to apheresis;
   8. Idelalisib (PI3Kδ kinase inhibitor) within 2 d prior to apheresis;
   9. DLI within 6 weeks prior to apheresis;
   10. Radiotherapy within 6 weeks prior to apheresis - progressive disease at radiotherapy site, or PET positive lesion at other non-radiotherapy site is eligible;
4. Patients previously received CAR-T cell therapy, the products that have same indication and have beenlisted in China are eligible;
5. Patients who have previously received allogeneic hematopoietic stem cell transplantation (allo-HSCT) within 3 mouths.
6. Patients with acute graft-versus-host disease (GVHD) or moderate-tosevere chronic GVHD within 4 weeks before screening.
7. Active systemic autoimmune disease.
8. Known infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus (HbsAg positive) or hepatitis C virus (anti- HCV positive).
9. Patients with active infections at screening.
10. History of cardiovascular disease.
11. Pregnant or nursing women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
【Phase I】Maximum Tolerated Dose (MTD), Dose Limiting Toxicity (DLT) and Recommended Phase II Dose (RP2D) | 28 days
  Determine the MTD and DLT of HY004 in the Treatment and recommend the dose for Phase II study.
【Phase II】Overall Remission Rate (ORR), which includes Complete Remission (CR) and Partial Remission (PR) | 3 months
  Efficacy of HY004 as measured by ORR at 3 months after HY004 Cell Injection infusion, which includes CR and PR.

SECONDARY OUTCOMES:
【Phase I】Overall Remission Rate (ORR), which includes Complete Remission (CR) and Partial Remission (PR) | 3 months
  Efficacy of HY004 as measured by ORR at 3 months after HY004 Cell Injection infusion, which includes CR and PR.
Safety of CNCT19 therapy: CTCAE v5.0 | 24 months
  Safety measures include adverse events as assessed by CTCAE v5.0.
Complete Remission Rate (CRR) | 3 months
  Efficacy of HY004 as measured by CR at 3 months after HY004 Cell Injection infusion.
ORR（CR+PR）/CRR | 28 days
  Efficacy of HY004 as measured by ORR/CRR at 28 days after cell infusion.
ORR（CR+PR）/CRR | 6 months
  Efficacy of HY004 as measured by ORR/CRR at 6 months after cell infusion.
Best Overall Response (BOR) | 24 mouths
  The best overall response after HY004 infusion.
Duration of Remission (DOR) | 24 mouths
  DOR means the duration from reaching the response (e.g., CR or PR) criteria of the therapy to the first, clearly defined progressive disease, or death for disease under investigation.
Progression-free survival (PFS) | 24 mouths
  PFS means duration from the HY004 Cell Injection infusion to progression of lymphoma, or death for any reason.
Event-free survival (EFS) | 24 mouths
  EFS means duration from the HY004 Cell Injection infusion to progression of lymphoma, start of new anti-cancer treatment, relapse, death of any cause or discontinued due to any adverse events.
Overall survival (OS) | 24 mouths
  OS is defined as the time from the signing of informed consent form to the date of the last survival follow-up or death due to any cause.

OTHER OUTCOMES:
In vivo cellular Pharmacokinetic (PK) profile of HY004. | 24 mouths
  To characterize the in vivo cellular pharmacokinetic (PK) profile (levels, persistence, trafficking) of HY004 cells in blood by quantitative polymerase chain reaction(qPCR) and Flow Cytometry.
In vivo cellular pharmacodynamics (PD) profile of HY004. | 3 mouths
  To characterize the concentration of cytokines ,including Interleukin-6(IL-6) at least in Serum.
Prevalence and incidence of humoral immunogenicity to HY004. | 24 mouths
  To characterize the concentration of anti-drug antibodies

IPD SHARING:
Plan to Share IPD: No